CLINICAL TRIAL: NCT01058525
Title: Influence of Ultrasonographic Hydro-dissection With Glucose 5% Solution on Median Nerve Block Efficiency: a Prospective and Randomized Study
Brief Title: Influence of Ultrasonographic Hydro-dissection With Glucose 5% on Nerve Block Efficiency
Acronym: Hydro-Echo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009/27
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Nerve Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- nerve block (Active Comparator): median nerve block (6 ml lidocaine 1.5 % with adrenalin 1:200000)
  Interventions: Procedure: median nerve block
- median nerve block after hydro-dissection (Experimental): median nerve block (6 ml lidocaine 1.5 % with adrenalin 1:200000) after hydro-dissection (glucose 5% solution)
  Interventions: Procedure: median nerve block after hydro-dissection

INTERVENTIONS:
Procedure: median nerve block — median nerve block performed using ultrasound guidance
  Arms: nerve block
Procedure: median nerve block after hydro-dissection — median nerve block performed after hydro-dissection (glucose 5% solution), both using ultrasound guidance
  Arms: median nerve block after hydro-dissection

SUMMARY:
The real-time visualization of a needle and nerve during an ultrasound-guided nerve block can be challenging. These difficulties may partly explain the systemic complications of local anesthetics under ultrasound. Injection of small amounts of a solution around the anesthetized nerve (hydro-dissection) has been proposed to enhance contrast outlining its borders and also to improve the visualization of the needle tip. The glucose solution 5% solution is interesting because it allows, unlike saline, to maintain the motor response with neurostimulation. The hydro-dissection can be particularly useful when one suspect hypoechoic vessels near the nerve to be anesthetized. Thereby, the nerve well demarcated and separated from the vessels, injection of local anesthetic is performed in the circumferential diffusion space (like a small pocket) without redirecting needle.

The influence of this hydro-dissection on the nerve block efficiency is unknown. The nerve block quality can be improved because the entire anesthetic is injected in contact with the nerve, but it can also be reduced due to the dilution of the local anesthetic by the glucose solution.

In this randomized study, the investigators test the hypothesis that hydro-dissection does not alter the nerve block onset time.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with an ASA physical status I-II scheduled for elective ambulatory surgery of the hand or wrist involving the median nerve

Exclusion Criteria:

* Patients with type 1 or 2 diabetes mellitus,
* History of clinical or laboratory evidence of abnormal bleeding,
* Infection at the injection site,
* Allergy to local anesthetic,
* Preexisting central or peripheral muscular or neurological disease (for example: carpal tunnel syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Onset time of sensory blockade (light touch test: total loss of sensation at the two distal phalanges of index) | 30 minutes after injection

SECONDARY OUTCOMES:
Onset time of sensory blockade (cold test at index finger and thenar eminence) | 30 minutes after injection
Onset time (light touch test at thenar eminence) | 30 minutes after injection
Onset time for motor blockade | 30 minutes after injection
Success rate (% of patients with total light touch block at index finger within 30 min evaluation period) | 30 minutes after injection
Successful surgical anesthesia | 30 minutes after injection
Duration of nerve blockade | 12 hours
Nerve block complication | one month
Duration of the puncture procedure | 30 minutes after the beginning of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, Study Chair — Hôpital Foch
Locations (1):
- Hôpital Privé de l'Ouest Parisien, Trappes, France

REFERENCES:
- [Derived] Dufour E, Donat N, Jaziri S, Kurdi O, Couturier C, Dreyfus JF, Fischler M. Ultrasound-guided perineural circumferential median nerve block with and without prior dextrose 5% hydrodissection: a prospective randomized double-blinded noninferiority trial. Anesth Analg. 2012 Sep;115(3):728-33. doi: 10.1213/ANE.0b013e31825fa37d. Epub 2012 Jun 28. PMID 22745114